CLINICAL TRIAL: NCT02947737
Title: Investigating the Effects of Amniotic Membrane on Donor Site Healing and Postoperative Pain
Brief Title: Amniotic Membrane for Donor Site Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Rachael Williams, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00088758
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Burns
Keywords: Skin graft
MeSH Terms: conditions — Burns | interventions — Biological Dressings; Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amniotic membrane dressing (Experimental): One donor site per study participant will be covered with an amniotic membrane dressing.
  Interventions: Other: Amniotic membrane dressing
- Gentamicin and xeroform dressing (Active Comparator): One donor site per study participant will be covered with a gentamicin and xeroform dressing.
  Interventions: Other: Gentamicin and xeroform dressing

INTERVENTIONS:
Other: Amniotic membrane dressing — We will place an amniotic membrane dressing on the donor site
  Arms: Amniotic membrane dressing
Other: Gentamicin and xeroform dressing — We will place xeroform, gentamicin and telfa on the donor site
  Arms: Gentamicin and xeroform dressing

SUMMARY:
The purpose of this study is to compare the effectiveness of applying amniotic membrane dressings compared to gentamicin and xeroform dressings to donor sites for skin grafts. This study will enroll ten participants who undergoing a split thickness skin graft procedure with two or more donor sites. The amniotic membrane will be applied to one donor site and a dressing of xeroform and gentamicin will be applied to another other donor site. Each participant will receive both types of dressing and will serve as their own control. Postoperative follow up will follow standard of care, regardless of the dressing type. Dressings will be removed on postoperative day 4 and participants will return to be re-examined one week after being discharged from the hospital.

DETAILED DESCRIPTION:
The use of amniotic membrane in the treatment of wounds has been employed for almost 100 years, with reports of it being used in skin grafting for burns and ulcers in 1913. This study will investigate the use of amniotic membrane as a donor site dressing (the area where skin is removed to be transplanted to the recipient site). Donor sites are often a significant cause of postoperative pain for patients who have undergone skin grafts. Furthermore, donor sites that fail to re-epithelialize or scar may require additional excision and skin grafting on the donor site itself. There is a paucity of literature in the United States regarding the use of amniotic membrane as a donor site dressing, however, studies from other countries have demonstrated an increase in patient comfort and a faster time to re-epithelialization. Inherent to amniotic membrane that makes it an ideal dressing include the presence of extracellular matrix components create integrity, epithelial cells participate in the healing process, and defensins confer antibacterial properties. MiMedx produces AmnioFix® which is a dehydrated preserved amniotic membrane that will be used in the dressing of our donor sites in contrast to gentamicin and xeroform based dressings. This study will see if patients have improved cosmetic outcomes, less postoperative pain and a faster time to re-epithelialization at the donor site treated with amniotic membrane compared to the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* undergoing a split thickness skin graft procedure with two or more donor sites

Exclusion Criteria:

* less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain | Postoperative days 1, 2 and 5
  Participants will report their pain level for each donor site as a numeric score from 1 to 10.
Change in re-epithelialization | Postoperative days 2 and 5
  The percent of re-epithelialization for each donor site will be evaluated by burn unit surgeons on postoperative days 2 and 5.
Comparison of scarring between donor sites | Postoperative day 5
  Scarring on postoperative day 5 will be evaluated by burn unit surgeons
Comparison of hypopigmentation between donor sites | Postoperative day 5
  Hypopigmentation on postoperative day 5 will be evaluated by burn unit surgeons.

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Williams, MD, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States